CLINICAL TRIAL: NCT05189691
Title: The Effect of Walking Exercises Performed Using Behavior Change Model on Symptom Severity and Quality of Life in Patients With Atrial Fibrillation: A Randomized Controlled Trial
Brief Title: The Effect of Walking Exercises in Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Ayse Ucar, Lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21149003
Record Dates: First submitted 2021-12-05; First posted 2022-01-12 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation; Quality of Life; Symptoms and Signs
Keywords: atrial fibrillation; behavior modification model (COM-B); walking exercise; symptom severity; quality of life
MeSH Terms: conditions — Atrial Fibrillation; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- behavior change and walking exercise (Experimental): A nurse-led interview will be held about the health benefits of lifestyle change and regular physical activity, which are effective in all CV diseases.Initially starting with 10-15 minutes of physical activity, it will continue until it reaches a duration of 30 or 60 minutes, 3 times a week. The goal is to exceed the previous number of steps each time. A pedometer will be used to ensure regular follow-up and control, and the number of steps will be marked on the walking tracking chart. They will be told how to keep a record after each exercise. A weekly phone call will be made to motivate the patient and the researcher will be informed that they can call.Blood pressure measurement, BMI, Toronto AF Symptom Severity Scale, Short Form 36 (SF-36) scales and continuously recorded step counts will be evaluated at week 0, 4 and at the end of week 12.
  Interventions: Behavioral: walking exercise
- behavior change (No Intervention): A nurse-led interview will be held about the health benefits of lifestyle change and regular physical activity, which are effective in all CV diseases.Blood pressure measurement, BMI, Toronto AF Symptom Severity Scale and Short Form 36 (SF-36) scales will be evaluated at week 0, 4 and at the end of week 12.

INTERVENTIONS:
Behavioral: walking exercise — Initially starting with 10-15 minutes of physical activity, it will continue until it reaches a duration of 30 or 60 minutes, 3 times a week. The goal is to exceed the previous number of steps each time. If they feel fatigue or palpitations during the day, they can do their exercises the next day. If there are complaints of shortness of breath/shortness of breath, chest pain, palpitation during walking, he should take a break from walking and rest. A pedometer will be used to ensure regular follow-up and control, and the number of steps will be marked on the walking tracking chart. They will be told how to keep a record after each exercise. A weekly phone call will be made to motivate the patient and the researcher will be informed that they can call.
  Other Names: behavior change
  Arms: behavior change and walking exercise

SUMMARY:
This research will be carried out to determine the effect of walking exercises performed using a behavioral change model on symptom severity and quality of life in patients with Atrial Fibrillation.

DETAILED DESCRIPTION:
Unique value of the project: Atrial fibrillation (AF) is one of the cardiovascular (CV) problems with a significant disease burden associated with stroke, for both patients and healthcare providers worldwide. Worldwide, AF is the most common sustained cardiac arrhythmia in adults, with an estimated prevalence ranging between 2% and 4%. In our country, this rate is between 1.25% and 1.4%. Patients with AF have a significantly poorer health-related quality of life compared with both healthy individuals and those with other cardiovascular diseases. This has been reported to be due to the various symptoms that AF patients may experience, such as fatigue, palpitations, dyspnea, sleep difficulties, chest discomfort, and psychosocial distress, as well as anxiety related to treatments and potential complications. An important step in AF management in AF guidelines is the optimization of cardiovascular and comorbidity and the identification and management of comorbidities, cardiometabolic risk factors, and unhealthy lifestyle factors to achieve this. As a lifestyle change in AF management, modifiable factors that may pose a risk for all cardiovascular disease (CVD) and AF are emphasized. Obesity and effective weight control, blood pressure control, increased physical activity and implementation strategies to achieve other risk factor modification, care pathways and education are the topics covered in this context. Exercise is a modifiable lifestyle factor that can affect AF risk both before and after AF onset. However, the recommended frequency, duration, and intensity of exercise in particular affect AF patients in different ways. The need to provide additional benefit to the current medical treatment is increasing day by day, and it is generally accepted that this benefit can only be achieved by changing the lifestyle of individuals and the continuity of this behavior change. The recommendation of the guidelines for AF patients is that they should focus on lifestyle change. Again in the guidelines, the success of nurse-led studies in AF patient management is a remarkable finding. According to the behavior change model, by evaluating the abilities and opportunities of the individual, by providing motivation under the leadership of the nurse, behavioral change can be targeted in the individual and self-monitoring and self-management of the individual can be realized in the long term. Regulating nutrition and weight control, reducing and managing alcohol intake, controlling high blood pressure and increasing physical activity, and maintaining behavior change with the support and motivation of nurses will be beneficial in AF patients to make lifestyle changes in AF patients. Although there are studies on physical activity in the AF patient group in the literature, no similar study has been found in our country. In addition, studies are insufficient in terms of creating evidence, and it is emphasized that more studies are needed. For this purpose, it is planned to conduct a nurse-led intervention study based on a behavioral change model in order to encourage physical activity, which is one of the subtitles of lifestyle change, in adults with AF.

Method: The project was planned as a prospective, single-blind, randomized controlled experimental type. The research will be carried out in Konya Necmettin Erbakan University Meram Medical Faculty Hospital Cardiology Department between March - October 2022. In determining the sample size, based on the studies in the literature, considering possible losses, and with 95% confidence and 80% test power, the minimum number of samples in each group was determined as 39 and a total of 78. In the collection of study data, the application steps of the Behavior Change Model and Behavior Change Wheel will be discussed first. Patient identification form, Short Form 36 (SF 36), University of Toronto Atrial Fibrillation Severity Scale (AFSS), Walk Tracking Chart and Pedometer (Pedometer) will be used as data collection tools.

Management: Data will be collected by the assistant researcher at the beginning of the study, at the 4th and 12th weeks, in the new service building of the Necmettin Erbakan University Meram Medical Faculty Hospital, in the echocardiography laboratory doctor's room.

In the preliminary application of the research, a questionnaire will be applied to 10 participants. In addition, to test the step counting accuracy of the pedometers according to the walking style, 5 participants will be visually counted and confirmed by the assistant researcher while walking at their own pace in the closed corridor.

Application

* When the implementation phase of the research begins, the purpose of the research will be explained and written/verbal consent will be obtained by interviewing individuals with AF sent by a cardiology specialist at the Necmettin Erbakan University Meram Medical Faculty Hospital Cardiology Clinic or outpatient clinic. Consent will be taken in the echocardiography laboratory doctor's room, where data are collected. Individuals who agree to participate in the research will be evaluated in terms of inclusion and exclusion criteria.
* As part of current clinical practice, all participants' blood pressure (BP), height and weight will be measured by the assistant researcher at study initiation. The patient identification form, the Toronto AF Symptom Severity Scale and Short Form 36 (SF-36) will be evaluated by interview method at baseline.
* Afterwards, an interview will be held by the assistant researcher about the lifestyle changes that are effective in all CV diseases and the health benefits of regular physical activity. Participants will be informed about the study and their written consent will be obtained.
* Participants included in the intervention group during the implementation phase of the study will be told that physical activity will start with 10-15 minutes initially, and then continue until participants reach a duration of 30 or 60 minutes, 3 times a week. Participants will be instructed that the goal is to exceed the previous number of steps each time.
* Participants will be informed that if participants feel fatigue or palpitations throughout the day, participants can exercise the next day.
* If participants have trouble/shortness of breath, chest pain, palpitation complaints during walking, he/she will be told to take a break from walking and rest. In addition to the controls of the participants with ongoing symptoms, the study will be carried out under the supervision of a cardiologist throughout the study.
* In order to ensure regular follow-up and control of the participants, a pedometer will be given and an explanation will be given about its use, and the participants will be asked to mark them on the walking tracking chart. After each exercise, the assistant researcher will explain to the participants how to keep a record.
* The initial step count value will be recorded as the number of steps recorded on the first day the participant used the pedometer.
* Participants will be instructed to put on the pedometer before walking and not to take it off during the walk. It will be emphasized that rhythmic walking is important for the pedometer to count correctly.
* Phone calls will be made once a week in order to motivate the participants, and participants will be informed that participants can call the assistant researcher for consultation when needed.
* Participants in the control group will receive standard clinical care.
* BP measurement, body mass index (BMI), Toronto AF Symptom Severity Scale and Short Form 36 (SF-36) scales will be evaluated by the assistant researcher at the 4th week and at the end of the 12th week in the experimental and control groups.
* In addition, the number of steps recorded continuously in the experimental group will be evaluated for analysis, taking into account the last measurements of the 4th and 12th weeks.

Widespread effect: Studies have shown that physical activity increases the quality of life, exercise capacity, heart rate control, peak maximum oxygen consumption (VO2 max) value, and reduces symptoms in AF patients. General population studies show that mild to moderate physical activity is primarily and secondarily protective against AF. Given the well-defined effects of prolonged exercise on the risk of AF, it has been reported that the optimal exercise interval for adults may be 20 minutes of aerobics, walking or cycling, 3 to 5 times per week. However, achieving less than recommended levels of physical activity was associated with a reduced risk of mortality compared to inactive patients, suggesting that even below recommended levels of physical activity, it is better than nothing for secondary prevention of AF.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-75
* Volunteer
* Sign the informed consent form
* Diagnosed with AF
* Speak and understand Turkish

Exclusion Criteria:

* Does not sign the informed consent form
* Not being literate
* Having cognitive and affective problems (vision, hearing impairment, delirium, dementia, depression, schizophrenia, bipolar disorder, etc.)
* Having had a myocardial infarction in the last month,
* Unstable clinical condition (uncontrolled cardiac arrhythmia, symptomatic severe aortic stenosis or other valvular disease, decompensated symptomatic heart failure and acute myocarditis or pericarditis),
* Presence of disability that will prevent physical activity (Orthopedic reasons or other disabilities).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation Symptom Severity | 4 weeks after the first assessment
  As a result of behavioral change, there will be a relationship between walking exercises measured with a pedometer and the University of Toronto Atrial Fibrillation Severity Scale (AFSS).Two separate scores are calculated on the scale: Atrial Fibrillation Burden and Atrial Fibrillation symptom severity:
  Total Atrial Fibrillation Burden = Atrial Fibrillation frequency + Atrial Fibrillation duration + Atrial Fibrillation severity. Each of the 3 measurements contributes equally to the Total Atrial Fibrillation load, each scoring a score of 1-10 and thus the total Atrial Fibrillation load will score a score of 3-30. Higher scores indicate greater Atrial Fibrillation burden.
  Atrial Fibrillation symptom severity: The scores obtained from the questions in Part C are summed (between 0-5) to calculate the total score. The total score is between 0-35. This score is the symptom severity score, and a higher score indicates an increased Atrial Fibrillation symptom severity.
Quality of Life with SF-36 | 4 weeks after the first assessment
  As a result of behavioral change, there will be a relationship between walking exercises measured by pedometer and RAND- 36 Item Short Form Survey Instrument (SF 36) score. SF-36 is a 36-item self-assessment scale consisting of eight subscales. This scale includes physical function (10 items), role limitations (physical (4 items)) and emotional problems (3 items), pain (2 items), vitality (4 items), social function (2 items), mental health (5 items)) and general health (5 items) subscales.
  Each subscale is scored between 0-100, with "0" the lowest and "100" the best quality of life.
Atrial Fibrillation Symptom Severity | 12 weeks after the first assessment
  As a result of behavioral change, there will be a relationship between walking exercises measured with a pedometer and the University of Toronto Atrial Fibrillation Severity Scale (AFSS).Two separate scores are calculated on the scale: Atrial Fibrillation Burden and Atrial Fibrillation symptom severity:
  Total Atrial Fibrillation Burden = Atrial Fibrillation frequency + Atrial Fibrillation duration + Atrial Fibrillation severity. Each of the 3 measurements contributes equally to the Total Atrial Fibrillation load, each scoring a score of 1-10 and thus the total Atrial Fibrillation load will score a score of 3-30. Higher scores indicate greater Atrial Fibrillation burden.
  Atrial Fibrillation symptom severity: The scores obtained from the questions in Part C are summed (between 0-5) to calculate the total score. The total score is between 0-35. This score is the symptom severity score, and a higher score indicates an increased Atrial Fibrillation symptom severity.
Quality of Life with SF-36 | 12 weeks after the first assessment
  As a result of behavioral change, there will be a relationship between walking exercises measured by pedometer and RAND- 36 Item Short Form Survey Instrument (SF 36) score. SF-36 is a 36-item self-assessment scale consisting of eight subscales. This scale includes physical function (10 items), role limitations (physical (4 items)) and emotional problems (3 items), pain (2 items), vitality (4 items), social function (2 items), mental health (5 items)) and general health (5 items) subscales.
  Each subscale is scored between 0-100, with "0" the lowest and "100" the best quality of life.

SECONDARY OUTCOMES:
Blood Pressure | 4 weeks after the first assessment
  As a result of behavioral change, there will be a relationship between walking exercises measured with a pedometer and systolic blood pressure and diastolic blood pressure.
BMI | 4 weeks after the first assessment
  As a result of behavioral change, there will be a relationship between walking exercises measured with a pedometer and BMI.
Blood Pressure | 12 weeks after the first assessment
  As a result of behavioral change, there will be a relationship between walking exercises measured with a pedometer and systolic blood pressure and diastolic blood pressure.
BMI | 12 weeks after the first assessment
  As a result of behavioral change, there will be a relationship between walking exercises measured with a pedometer and BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Selda ARSLAN, Phd, Study Director — Necmettin Erbakan University Faculty of Nursing; Ayşe Uçar, MSC, Principal Investigator — Necmettin Erbakan University Faculty of Nursing
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No